CLINICAL TRIAL: NCT00487903
Title: A Phase 2 Trial of PB127 Myocardial Perfusion Echocardiography to Evaluate and Optimize Additional Ultrasound Imaging Systems
Brief Title: Evaluation and Optimization of PB127 Myocardial Perfusion Echocardiography on Ultrasound Systems
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinued PB127 development program for business reasons
Sponsor: Point Biomedical (Industry)
Responsible Party: Tom Ottoboni, PhD/Chief Operating Officer, Point Biomedical Corp.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 127-015
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2008-07-03 (Estimated); Status verified 2008-07

CONDITIONS: Coronary Artery Disease; Healthy
Keywords: Coronary Artery Disease; Echocardiogram; Contrast; Perfusion; Ultrasound; Normal volunteers
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PB127 for Injectable Suspension — 0.062 mg/kg continuous IV (100-250 mL/hr) during echocardiogram, single dose, infusion not to exceed 60 minutes.
  Other Names: CARDIOsphere®

SUMMARY:
The purpose of this clinical trial is to evaluate various commercially available ultrasound systems and to identify imaging parameters to be used with these systems (along with the contrast agent PB127) as well as to further evaluate the safety of PB127.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women

1. Normal volunteers (18 30 years old), with no history of CAD
2. Patients (≥ 18 years old) with known or suspected CAD, scheduled for or undergone clinically indicated coronary angiography within 28 days prior to or following Study Day 1

Exclusion Criteria:

1. Unable to provide written informed consent
2. Women who are pregnant or lactating
3. Known hypersensitivity or known contraindication to:

   1. Dipyridamole
   2. Ultrasound contrast agents (including PB127 and excipients)
   3. Blood, blood products, albumin, egg whites, or protein
4. Use of caffeine or xanthine containing products within the 24 hours prior to PB127 administration on Study Day 1
5. Previous exposure to PB127
6. Inadequate echocardiographic windows
7. Heart transplant
8. Known right to left shunt, including atrial septal defect
9. History of CABG
10. Current uncontrolled ventricular tachycardia, atrial fibrillation, atrial tachycardia, or atrial flutter
11. Pacemaker or defibrillator
12. Unstable angina grade CCS Class IV severity with ongoing symptoms and/or ongoing infusion of IV nitroglycerin
13. Second degree or greater heart block
14. Hypertension (SPB >200 and/or DBP >110 mmHg on two consecutive readings within 1 hour prior to PB127 administration)
15. Hypotension (SPB <90 mmHg on two consecutive readings within 1 hour prior to PB127 administration)
16. Severe aortic stenosis (>100 mmHg peak transvalvar gradient or <0.6 cm2 estimated valve area)
17. Pulmonary edema within the 7 days prior to Study Day 1
18. Resting oxygen saturation of less than 90%
19. Q wave MI within the 7 days prior to Study Day 1
20. PTCA within the 28 days prior to Study Day 1
21. Chronic obstructive pulmonary disease or bronchospastic airway disease which, in the opinion of the Investigator, is significant enough to contraindicate dipyridamole
22. Known history of severe pulmonary hypertension characterized by estimated pulmonary artery systolic pressure of >50 mmHg
23. Liver disease, characterized by or including one or more of the following

    1. Elevated total bilirubin >upper limit of normal
    2. Currently elevated hepatic enzymes >3X upper limit of normal
24. Medical conditions or other circumstances that would significantly decrease the chances of obtaining reliable data or achieving the study objectives (i.e., drug dependence, psychiatric disorder, dementia, or associated illness); extenuating circumstances or medical conditions that make it unlikely that a patient can complete the clinical trial or follow up evaluations; or other reasons for expected poor compliance with the clinical investigator's instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Determination of optimal machine settings and imaging parameters for myocardial perfusion for a variety of ultrasound imaging systems to be used in upcoming clinical trials | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ehlgen, MD, PhD, Study Director — POINT Biomedical Corp.
Locations (3):
- United States (3):
  - Midwest Cardiology Associates, Overland Park, Kansas
  - Duke University Medical Center, Durham, North Carolina
  - Baylor Research Institute, Dallas, Texas